CLINICAL TRIAL: NCT05810961
Title: A Multicenter, Randomized, Double-blinded, Placebo-controlled, Proof-of-Concept Study to Evaluate the Efficacy and Safety of Efgartigimod in Chinese Patients with Primary Membranous Nephropathy
Brief Title: A Study to Assess Effectiveness and Safety of Efgartigimod in Chinese Patients with Primary Membranous Nephropathy (ZL-1103-014)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: argenx (Industry)
Collaborators: Zai Lab Pty. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ARGX-113-2203
Record Dates: First submitted 2023-03-29; First posted 2023-04-13 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Membranous Nephropathy
Keywords: kidney disease; Glomerulonephritis membranous; Urologic disease; glomerulonephritis
MeSH Terms: conditions — Glomerulonephritis, Membranous; Kidney Diseases; Urologic Diseases; Glomerulonephritis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- efgartigimod IV (Experimental): patients receiving infusions of efgartigimod
  Interventions: Biological: efgartigimod IV
- placebo (Experimental): patients receiving infusions of placebo
  Interventions: Other: placebo

INTERVENTIONS:
Biological: efgartigimod IV — infusion of efgartigimod
  Arms: efgartigimod IV
Other: placebo — infusion of placebo
  Arms: placebo

SUMMARY:
To evaluate the efficacy and safety of efgartigimod IV in Chinese patients with primary membranous nephropathy (pMN).

DETAILED DESCRIPTION:
To evaluate the efficacy and safety of efgartigimod IV in Chinese patients with primary membranous nephropathy (pMN).The study comprises a maximum 4-week screening period, a 24-week treatment period, and an 8-week follow-up period

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥18 years when signing the informed consent form (ICF)
* Capable of providing signed informed consent and complying with protocol requirements
* Diagnosis of idiopathic (primary) MN confirmed by renal biopsy within 24 months before randomization. A renal biopsy may be taken at any time during the screening period to confirm the diagnosis of MN for participant eligibility, if the most recent biopsy was performed greater than 24 months before randomization
* Receiving stable dose at maximum tolerated or allowed dose of ACEi and/or ARB for at least 12 weeks before randomization
* Agree to use contraceptives consistent with local regulations. Full inclusion criteria can be found in the protocol

Exclusion Criteria:

* Active or chronic infection requiring treatment
* Diagnostic renal biopsy showing evidence of crescent formation in glomeruli, suggestive of an alternative or additional diagnosis to pMN; evidence on renal biopsy of >50% interstitial fibrosis/tubular atrophy in the cortical area
* History of malignancy unless deemed cured by adequate treatment with no evidence of recurrence for ≥3 years before randomization.
* Any evidence of diabetic glomerulopathy on renal biopsy that is:

Greater than Class I diabetic glomerulopathy, or Class I diabetic glomerulopathy with a history of poor diabetic control (eg, HbA1c ≥9.0%) since time of biopsy

* Currently on renal dialysis or expected to require dialysis during study period
* Previous kidney transplantation or planned transplantation during study period
* Any other known autoimmune disease that, requires systemic immunosuppressive treatments, or in the opinion of the investigator, would interfere with an accurate assessment of clinical symptoms of pMN or put the participant at undue risk
* Clinical evidence of other significant or uncontrolled serious diseases (ie, cardiovascular, pulmonary, hematologic, gastrointestinal, hepatic, renal, neurological), have had a recent major surgery, or have any other condition, that in the opinion of the investigator, could confound the results of the study or put the participant at undue risk
* Use of complementary therapies, including Traditional Chinese Medicine, herbs, or procedures (eg, acupuncture) within 4 weeks before randomization that can potentially interfere with the efficacy and safety of participants as assessed by the investigator
* Received live/live-attenuated vaccine within 28 days before randomization. The receipt of any inactivated, subunit, polysaccharide, or conjugate vaccine at any time before screenings is not considered exclusionary. It is recommended that participants are up to date with vaccination before the first dose of IMP
* Previously participated in a clinical study with efgartigimod
* SARS-CoV-2 positive test at screening. The test is required regardless of whether the participant has been vaccinated
* Known hypersensitivity or contraindication to efgartigimod, or any excipient of the IMP
* In the opinion of the investigator, current or history of (ie, within 12 months of randomization) alcohol, drug, or medication abuse
* Pregnant or lactating females and those who intend to become pregnant during study participation
* Any conditions or circumstances that in the opinion of the investigator may make the participant unsuitable for the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2023-02-20 (Actual); Primary Completion 2024-08-05 (Actual); Study Completion 2024-08-05 (Actual)

PRIMARY OUTCOMES:
Change from baseline to week 24 in urine protein creatinine ratio (UPCR) in anti- PLA2R antibody (Ab) seropositive population | up to 24 weeks

SECONDARY OUTCOMES:
Change from baseline to week 24 in urine protein creatinine ratio (UPCR) in overall population | up to 24 weeks
Proportion of participants achieving complete remission (CR), defined as proteinuria ≤0.3g/24-hour and serum albumin ≥3.5g/dL, at week 24 in overall population and anti-PLA2R Ab seropositive population | up to 24 weeks
Time to complete remission (CR) in overall population and anti-PLA2R Ab seropositive population | up to 32 weeks
Proportion of participants achieving partial remission (PR), defined as ≥50% reduction in proteinuria from baseline AND final proteinuria between 0.3 to 3.5g/24-hour, at week 24 in overall population and anti-PLA2R Ab seropositive population | up to 24 weeks
Time to partial remission (PR) in overall population and anti-PLA2R Ab seropositive population | up to 32 weeks
Change from baseline to week 24 in anti-PLA2R Ab in anti-PLA2R Ab seropositive population | up to 24 weeks
Change from baseline to week 24 in serum albumin in overall population and anti-PLA2R Ab seropositive population | up to 24 weeks
Change from baseline to week 24 in estimated glomerular filtration rate (eGFR) in overall population and anti-PLA2R Ab seropositive population | up to 24 weeks
Treatment failure rate during treatment period in overall population and anti-PLA2R Ab seropositive population | up to 32 weeks
Incidence of relapse, defined as the development of nephrotic range proteinuria following CR or PR, ie, >3.5g/24-hour throughout the study in overall population and anti-PLA2R Ab seropositive population | up to 32 weeks
Efgartigimod serum concentration-time profile in overall population and anti-PLA2R Ab seropositive population | up to 32 weeks
changes from baseline in levels of total IgG | up to 32 weeks
Incidence of antidrug antibodies (ADA) against efgartigimod in overall population and anti-PLA2R Ab seropositive population | up to 32 weeks
Change from baseline in EQ5D-5L score in overall population and anti-PLA2R Ab seropositive population | up to 24 weeks
Change from baseline in PROMIS Short form v1.0 Fatigue-4a questionnaire in overall population and anti-PLA2R Ab seropositive population | up to 24 weeks

CONTACTS AND LOCATIONS:
Locations (31):
- China (31):
  - Peking University People's Hospital, Beijing
  - Hunan Provincial People's Hospital, Changsha
  - The Second Affiliated Hospital of Chongqing Medical University, Chongqing
  - Fujian Medical University Union Hospital, Fujian
  - Fuyang People's Hospital, Fuyang
  - Guangdong Provincial People's Hospital, Guangzhou
  - Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou
  - The First Affiliated Hospital, Sun Yat-sen University, Guanzhou
  - The First Affiliated Hospital, Zhejiang University, Hanzhou
  - The Second Hospital of Anhui Medical University, Hefei
  - The Affiliated Huaian No.1 People's Hospital of Nanjing Medical University, Huai'an
  - Shandong Provincial Hospital Affiliated to Shandong First Medical University, Jinan
  - Liu Zhou Works Hospital, Liuchow
  - The First Affiliated Hospital of Nanchang University, Nanchang
  - Jiangsu Province Hospital, Nanjing
  - Zhongda Hospital Southeast University, Nanjing
  - The People's Hospital of Guangxi Zhuang Autonomous Region, Nanning
  - Pingxiang People's Hospital, Pingxiang
  - Huashan Hospital Fudan University, Shanghai
  - Renji Hospital Shanghai Jiaotong University School of Medicine, Shanghai
  - ShengJing Hospital of China Medical University, Shenyang
  - Shenzhen People's Hospital, Shenzhen
  - The First Hospital of Hebei Medical University, Shijia Zhuang
  - The Second Hospital of Tianjin Medical University, Tianjin
  - Renmin Hospital of Wuhan University, Wuhan
  - Wuxi People's Hospital, Wuxi
  - Shaanxi Provincial Hospital of Chinese Medicine, Xi'an
  - The First Affiliated Hospital of Xiamen University, Xiamen
  - Xiamen Fifth Hospital, Xiamen
  - Henan Provincial People's Hospital, Zhengzhou
  - Zhuhai People's Hospital, Zhuhai

IPD SHARING:
Plan to Share IPD: No